CLINICAL TRIAL: NCT02015858
Title: Pain During Chest Tube Withdrawal: Evaluation Using Pan Monitor in Patients With or Without Epidural Anesthesia
Brief Title: Pain During Chest Tube Withdrawal: Evaluation Using Pan Monitor
Acronym: Pain Drain
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/22; 2013-A00612-43 (Other: ANSM)
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epidural analgesia: Postoperative patients with epidural analgesia
  Interventions: Procedure: Chest drain withdrawal; Device: Pain Monitor
- Oral analgesics: Postoperative patients with oral analgesics
  Interventions: Procedure: Chest drain withdrawal; Device: Pain Monitor

INTERVENTIONS:
Procedure: Chest drain withdrawal
Device: Pain Monitor
  Other Names: Measurement of Pain Monitor index

SUMMARY:
Pain evaluation remains a clinical problem. Pain Monitor allows pain evaluation using the measurement of skin conductance.

Withdrawal of chest tube can be painful and the purpose of the study was to compare auto-evaluation of pain (visual analogic scale) and the index measured by the Pain Monitor.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing removal of a chest tube after lung surgery,
* patients able to indicate the pain score.

Exclusion Criteria:

* pregnancy, lactation ,
* insulin-dependent diabetes with dysautonomia,
* central or peripheral neurological disease, agitation,
* inability to understand the protocol,
* inability to use the Pain Monitor: skin abnormalities at the site of measurement, pacemaker or implantable defibrillator, condition affecting the sympathetic nervous system, tremor of the extremities,
* contra-indication to oral morphine ,
* respiratory failure, severe hepatic insufficiency, intracranial hypertension, epilepsy associations
* recent administration of neostigmine or of atropine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain monitor evaluation of pain | 1 hour
  Comparison between Pain monitor index and auto-evaluation of pain (numerical scale from 0 -no pain- to 10 - maximal pain)

SECONDARY OUTCOMES:
Pain intensity | 1 hour
  Evolution of Pain monitor index and of auto-evaluation of pain (numerical scale from 0 -no pain- to 10 - maximal pain) during the chest tube withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, Study Chair — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, France